CLINICAL TRIAL: NCT05581420
Title: Oral Versus Intravenous Iron in IBD Patients With Anti-inflammatory Therapy
Acronym: OVI-IBD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: University Medical Center Groningen (Other); UMC Utrecht (Other); Rijnstate Hospital (Other); Erasmus Medical Center (Other); Sint Franciscus Gasthuis (Other); Adrz, Goes (Unknown); Medical Center Haaglanden (Other)
Responsible Party: Principal Investigator, Andrea E. van der Meulen - de Jong, MD, PhD, Principal Investigator, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL79363.058.21
Record Dates: First submitted 2022-08-17; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — ferrous fumarate; ferric carboxymaltose; Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral iron (Active Comparator): Ferrous fumarate 200mg daily for 4 weeks.
  Group A1 (Normal Hb at week 4):
  Ferrous fumarate 100mg daily for 12 weeks
  Group A2 (Abnormal Hb at week 4):
  Ferrous fumarate 200mg daily for 8 weeks
  Group A2 at week 12:
  Normal Hb: ferrous fumarate 100 mg daily till week 16 Abnormal Hb: intervention failure. End of study.
  Interventions: Drug: Ferrous fumarate
- IV Iron (Active Comparator): Dosage based on iron formulation and instructions according to recommended guidelines (weight of patient)
  Interventions: Drug: MonoFer

INTERVENTIONS:
Drug: Ferrous fumarate — Patients randomized in the oral group, will all be prescribed ferrous fumarate 200 mg d.d. for the first 4 weeks. Then, depending on their iron status, 100 mg d.d. for the following 12 weeks or 4 more weeks 200 mg d.d. followed by 4 weeks 100 mg d.d.. If iron levels are still too low after 12 weeks, the intervention has failed.
  Arms: Oral iron
Drug: MonoFer — Study patients will be treated with intravenous iron. The brand name of the iv iron is dependent on the hospital policy and the doses will be according to recommended guidelines (weight of patient). Iv iron is intramural medication without add-on status and needs infusion at daycare.
  Other Names: Ferinject; Cosmofer; Venofer
  Arms: IV Iron

SUMMARY:
Rationale: Iron deficiency anemia is the most common systemic manifestation of Inflammatory Bowel Diseases (IBD)-Crohn's disease and ulcerative colitis. Iron deficiency with or without anemia poses a diagnostic and therapeutic challenge due to chronic gastrointestinal blood loss and the inflammatory nature of IBD. Oral iron supplementation in active disease states is controversial. Hepcidin levels can be considered as the sum effect of all regulatory processes. Studies suggested that iron stores and hypoxia reduce hepcidin levels even in an inflammatory state. This is also reflected by a study which demonstrated low levels of hepcidin in patients with ferritin levels under 30μg/ml, regardless of disease activity or type. Furthermore, studies show that immunosuppressive medication decrease the level of hepcidin. This raises the question: is oral iron a viable alternative for patients under immunosuppressive treatment for active IBD? Objective: The hypothesis is that patients with mild to moderate IBD activity on immunosuppressive medication, show the same level of Hb increase after 12 weeks after either oral or iv iron supplementation, while the price of oral iron supplementation is significantly lower.

DETAILED DESCRIPTION:
Study design: multicenter, prospective randomized non-inferiority study. Study population: Patients with inflammatory bowel disease on immunosuppressive medication with iron deficiency anemia, with increased inflammation parameters, but without an elevated ferritin (<100 μg/L).

Intervention: 152 patients will be randomized to a treatment group with either low dose oral iron or iv iron supplementation.

Main study endpoints: Normalization of Hb concentration (> 7.3 mmol/L (females) or > 8.0 mmol/L (males)) from baseline to week 12 in both oral and iv iron supplementation group.

Patients will receive either oral or intravenous iron therapy. Both therapies will be given according to existing guidelines. Participation to this trial will not increase the frequency of regular follow-up visits for patients. Blood for study measurements will be drawn simultaneously as blood for standard care tests. In addition, three questionnaires will be sent out regarding the patient's quality of life, disease activity, and productivity impairment. Iron therapy and biomaterial acquisition do not increase patients' risk because patients would have to undergo the same tests for standard IBD-care and receive iron therapy outside of the study. The study will be directly beneficial to participating patients because patients will undergo treatment for iron deficiency. The findings might help to develop guidelines for personalized iron therapy in the IBD population.

ELIGIBILITY:
Inclusion Criteria:

* Established IBD diagnosis (Crohn's disease, ulcerative colitis, IBD-unclassified)
* Adults (≥18 years of age)
* Any single Hb level between 6,2 - 7,3 mmol/L (females) 6,2 - 8,0 mmol/L (males)
* Any single ferritin <100 μg/L and transferrin saturation <20% within 4 weeks of study inclusion
* CRP > 5 mg/L and / or fecal calprotectin > 150 within 4 weeks of randomization
* Patients on immunosuppressive medication (thiopurine, methotrexate, biologicals, JAK inhibitor) for at least 8 weeks or if prednisone, for at least 2 weeks
* Mild to moderate disease according to the treating physician; a Physician Global Assessment (PGA) score of 1 or 2
* Documented informed consent

Exclusion Criteria:

* Anemia due to reasons other than iron deficiency or chronic disease (e.g. hemoglobinopathy).
* Severe disease with a PGA score of 3
* IBD patients with a location of IBD at other places than ileum and / or colon (according to treating physician)
* Patients who are prescribed PPI
* Earlier significant side effect of oral iron or iv iron
* Folic acid deficiency (<2.5 μg/ml)
* Vitamin B12 deficiency (<150 mg/l)
* Patients can proceed with their regular diet, but during the study they cannot take supplements that contain iron. For example, commercial vitamins with iron or a well-known iron supplement Floradix®. Intake of said supplements must be stopped at the moment of inclusion.
* Documented history of bariatric surgery or gastric/duodenal resections due to benign or malignant pathologies
* Documented major operation (e.g., laparotomy) less than six weeks before inclusion
* Documented history of liver cirrhosis, heart failure, hemoglobinopathies, autoimmune hemolytic anemia, myelodysplastic syndrome, or chronic obstructive pulmonary disease (COPD)
* Documented history of recent treatment for a malignancy (excluding dermatological malignancies such as basal cell carcinoma or squamous cell carcinoma). Patients can be included if the treatment for malignancy has been finalized ≥6 months before the inclusion date.
* End-stage renal disease (impaired renal function, defined as eGFR <30 ml/min/1.73m2)
* Documented pregnancy or breastfeeding at the time of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Normalization of Hb concentration (> 7.3 mmol/L (females) or > 8.0 mmol/L (males)) from baseline to week 12 in both oral and iv iron supplementation group. | After 12 weeks
  Percentage of patients who achieved an adequate hematologic response (defined by Hb > 7.3 mmol/L (females) or > 8.0 mmol/L (males)) after 12 weeks

SECONDARY OUTCOMES:
Change in Hb levels | baseline, weeks 4, 12 and 16
  Change in Hb levels from baseline to weeks 4, 12, and 16 in both both oral and iv iron supplementation group.
percentage of participants with ferritin levels > 100 microg/l | after 4, 12 and 16 weeks
  Percentage of patients who achieve ferritin levels > 100 microg/l in both both oral and iv iron supplementation group.
Preference of patient for oral versus i.v. iron | at baseline and at week 16
  percentage of patients who prefer oral or i.v. iron supplementation
Change in Disease-specific Quality of life (IBDQ) | at week 16 in comparison with baseline
  Change in health related quality of life (measured by the sIBDQ) measuring physical, social, and emotional status (score 10-70, poor to good HRQoL) from baseline to week 16 in both both oral and iv iron supplementation group.
Change in overall/generic Quality of life (EQ-5D-5L) | at week 16 in comparison with baseline
  Change in overall/generic quality of life from baseline to week 16 in both oral and iv iron supplementation group. This is measured by the EQ-5D-5L generating a 5-digit number that describes the patient's health state and a VAS that can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Change in productivity cost (iPCQ) | at baseline and week 16
  Change in productivity cost (measured by the iPCQ) from baseline to week 16 in both both oral and iv iron supplementation group. To calculate the cost of productivity losses, volumes are multiplied by unit cost prices.
Change in medical consumption use (iMCQ) | at baseline and week 16
  Change in medical consumption use (measured by the iMCQ) from baseline to week 16 in both both oral and iv iron supplementation group. The costs of medical consumption are calculated by multiplying measured volumes of care by the cost per unit of care.
Therapy adherence measured with the modified MMAS-8 for patients in the oral iron group | at week 4, 8, 12 and at week 16 if patients still use iron according to the protocol
  Therapy adherence measured with the modified MMAS-8 for patients in the oral iron group. Scores of 8 points, <8 to >6 points and ≤6 points are considered to have high, medium and low adherence, respectively.
Correlation between response to iron therapy and disease activity | At week 4, 12 and 16
  he correlation of disease activity (evaluated by fecal calprotectin levels and c-reactive protein levels) and response to iron therapy in both oral and iv iron supplementation group.
Incidence of hypophosphatemia during iron therapy | At week 4, 12 and 16
  Percentage of patients who experienced hypophosphatemia throughout iron therapy in both oral and iv iron supplementation group.
Number of (serious) adverse events and adverse reactions according to MedDRA criteria. | From baseline until week 16
  Number of (serious) adverse events and adverse reactions according to MedDRA criteria throughout the study period.
Change in clinical disease activity | baseline, weeks 4, 12 and 16
  Change in clinical disease activity (measured by mobile Health Index (mHI) 0-24 for patients with Crohn's disease and 0-34 for patients with ulcerative colitis; higher scores indicate a more active disease) 16 in both oral and iv iron supplementation group from baseline to week 16.
Hepcidin - and soluble Transferrin Receptor (sTfR) - fecal calprotectin / CRP ratio | at baseline and week 12

CONTACTS AND LOCATIONS:
Overall Officials: A.E. van der Meulen - de Jong, MD, PhD, Principal Investigator — Leiden University Medical Centre
Locations (1):
- Leiden University Medical Centre, Leiden, South Holland, Netherlands